CLINICAL TRIAL: NCT04730713
Title: The Morphology and Parameter Estimation of Cranial Ultrasound Spectrum Based on Cerebral Artery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 202101009
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Intracranial Pressure Increase
Keywords: Transcranial Doppler（TCD）,Intracranial pressure(ICP)
MeSH Terms: conditions — Intracranial Hypertension | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Admitted to the center ICU due to neurosurgery, brain dysfunction and other neurological reasons: Aneurysmal subarachnoid hemorrhage (aSAH), traumatic brain injury (TBI), acute deficiency Blood stroke (AIS), acute cerebral hemorrhage (ICH), hypoxic ischemic encephalopathy (HIE), Sepsis-associated encephalopathy (SAE), intracranial tumor surgery; older than 18 years old, <85 Years old; patients who need lumbar puncture.
  Interventions: Device: The morphology and parameters of cranial ultrasound spectrum based on cerebral artery

INTERVENTIONS:
Device: The morphology and parameters of cranial ultrasound spectrum based on cerebral artery — Subjects who meet the standards will undergo a full-body examination and basic life after entering the ICU Sign evaluation and monitoring, mainly including nervous system specialist physical examination, multi-modal brain function testing, Respiratory system monitoring and management, hemodynamic monitoring, APACHE Ⅱ score, GCS score, and routine general circulation, respiratory management, sedation and analgesia management, temperature management, infiltration Pressure management, lumbar pressure measurement The included subjects were monitored for optic nerve sheath diameter, TCD/TCCD before and after lumbar puncture, and recorded spectrum morphology: normal, high resistance state, ischemic topic, congestion state, spasticity, nail wave/oscillating wave state, S1S2 fusion high point state, and recording at the same time Parameters: systolic flow rate (Vs) Shu Tensile blood flow velocity (Vd), average blood flow velocity (Vm), pulsatility index (PI), impedance Index (RI)
  Other Names: transcranial Doppler

SUMMARY:
1. Observe the changes of TCD/TCCD spectrum shape before and after lumbar puncture in patients with severe neurological disease.
2. Discuss the TCD/TCCD spectrum shape and parameters of cerebral arteries and neurocritical patients Correlation of intracranial pressure.

DETAILED DESCRIPTION:
After entering the ICU, the subjects who meet the standards will undergo a full-body physical examination and basic vital signs assessment and monitoring, which mainly include specialized examinations of the nervous system, multimodal brain function testing, respiratory system monitoring and management, hemodynamic monitoring, and APACHEⅡ Score, GCS score, and perform routine general circulation, breathing management, sedation and analgesia management, temperature management, osmotic pressure management, lumbar puncture pressure measurement

ELIGIBILITY:
Inclusion Criteria:

Aneurysmal subarachnoid hemorrhage (aSAH), traumatic brain injury (TBI), acute deficiency Blood stroke (AIS), acute cerebral hemorrhage (ICH), hypoxic ischemic encephalopathy (HIE), Sepsis-associated encephalopathy (SAE), intracranial tumor surgery; older than 18 years old, <85 Years old; patients who need lumbar puncture.

Exclusion Criteria:

1. Age <18 years old;
2. Pregnancy;
3. The condition of the temporal window is limited and the image cannot be obtained;
4. The frequency spectrum of bilateral cerebral arteries shows stenosis;
5. Patients with cerebral artery stenosis
6. Patients who have not obtained informed consent;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age over 18 years old, <85 Years old; patients who need lumbar puncture.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
The TCD/TCCD spectrum shape and parameters of cerebral arteries are related to the intracranial pressure of neurocritical patients | January 26, 2021 to December 30, 2022
  The change of TCD/TCCD spectrum shape can qualitatively evaluate ICP. The intracranial pressure is qualitatively determined by spectrum morphology to help clinicians quickly assess intracranial pressure and guide treatment. Accurately identify the normal shape of the spectrum, the state of high resistance, the state of ischemia, the state of congestion, the state of spasticity, the state of nail wave/oscillating wave, and the state of S1S2 fusion high tip. Discuss the correlation between spectrum shape and waist piercing ICP.

CONTACTS AND LOCATIONS:
Overall Officials: li na li na, PhD Tutor, Study Chair — Department of Critical Care Medicine, Central South University
Locations (1):
- medical Ethics committee of Xiangya Hospital Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No